CLINICAL TRIAL: NCT04401787
Title: Is There Better Oncological and Short Term Outcome for Laparoscopic Resection of Upper Rectal Carcinoma T1-4 N0-1 Over Laparoscopic Converted Cases in Obese Patients?
Brief Title: Converted Laparoscopic Resection of Upper Rectal Carcinoma T1-4 N0-1 in Obese Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Bassem Mohamed Sieda, Assistant professor of general surgery, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR-20780302-1
Record Dates: First submitted 2020-05-19; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Cancer, Rectum
Keywords: rectal cancer; laparoscopic resection; obesity
MeSH Terms: conditions — Rectal Neoplasms; Obesity | interventions — Adiposity

STUDY DESIGN:
Intervention Model Description: A prospective study included 191 patients, randomly allocated into two arms of the study, Arm I is open anterior resection (OAR), this is the control and arm II, The LAR. Only 156 analyzed.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic anterior resection (LAR) (Active Comparator): LAR group included 88 patients, 17 patients converted to open
  Interventions: Procedure: Anterior resection for upper rectal cancer in obese
- open anterior resection (Active Comparator): Open anterior resection for 56 patients
  Interventions: Procedure: Anterior resection for upper rectal cancer in obese

INTERVENTIONS:
Procedure: Anterior resection for upper rectal cancer in obese — Anterior resection for upper rectal cancer in obese

SUMMARY:
Background: laparoscopic resection (LAR) is a safe approach and widely used for rectal cancer after neoadjuvant chemo-radiotherapy, but short term and oncological outcome for converted cases to open surgery (cLAR), may be questioned in an obese patient.

Objective: validating the short-term and oncological outcomes after laparoscopic resection and after conversion to open surgery for upper rectal cancer in obese patients.

Patients and methods: A prospective study included 191 patients, randomly allocated into two arms of the study, Arm I is open anterior resection (OAR), this is the control and arm II, The LAR. Only 156 analyzed.

DETAILED DESCRIPTION:
Study design: A randomized control study assigned to involve obese patients with BMI 30 diagnosed with upper rectal carcinoma T1-4 N0-1, 181 patients assigned into two arms and operated in multi-centres in a tertiary hospitals.

Ethical approval and clinical registration: Our study was submitted, revised and finally permitted and approved by the Institutional Review Board of the Zagazig University hospital, faculty of medicine, holding number IR-20780302-1, and informed consent was obtained from all participants agreed to be involved. Study registered in ClinicalTrial.gove: ID: ………

Protocol and setting:

A study was done in the period from December 2016 to December 2019 and data registered after each procedure in our database system The controlled arm included patients underwent open anterior resection (OAR) for upper rectal carcinoma and divided into Ia, underwent OAR and IIa, included patients with cLAR, whereas Group II included patients underwent LAR.

Method of randomization:

Randomization was done via a computer-generated protocol, already designed and uploaded in our database, and the results were unlabeled and sealed into envelopes. These envelopes were opened in the operating room by the head-nurse and an assistant surgery specialist who was not engaged in the study

Inclusion criteria:

Obese patients with BMI ≥27 with operable upper rectal carcinoma staged T1-4 N0-1 based on colonoscopy, endo-rectal ultrasound, CT abdomen and pelvis and MRI abdomen Exclusion criteria BMI less than 27, According to AJCC TNM staging 7th edition, N2-3 patients were excluded, any evidence of inoperability whether distant metastasis or invasive tumours, Patients with synchronous colorectal tumours, synchronous liver metastasis obstructive symptomatic patients and patients with intraoperative tumour rupture or perforation, rectal tumours below peritoneal reflection.

There are 2 parameters prospectively assessed and registered in our database: First the clinical parameters, second is the onco-pathological parameter Clinical parameter included, operative basic demographic data (age, sex and BMI), peri-operative clinical variables ( operative time, intraoperative complication, completeness of TME, the feasibility of stapling, causes of conversion if there, postoperative (PO) short term outcome, Recovery, hospital stay, PO morbidity and bowel function.

The onco-pathological outcome included: tumour site, site and staging of tumour according to TNM- longitudinal and circumferential resection margin- LN involved (N) - loco-regional recurrence and recurrence-free survival.

Intervention methods The preoperative nCRT: our protocol according to a multidisciplinary tumour board committee, is to give a long course of neo-adjuvant chemo-radiotherapy for mid and lower rectal cancer but upper rectum, we give a 4 weeks course of CRT, 45 Gy with systemic 5-fluorouracil based regimen infusion. This is proposed for stage II-III not stage I.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients with BMI ≥27 with operable upper rectal carcinoma staged T1-4 N0-1 based on colonoscopy, endo-rectal ultrasound, CT abdomen and pelvis and MRI abdomen

Exclusion Criteria:

* BMI less than 27, According to AJCC TNM staging 7th edition, N2-3 patients were excluded, any evidence of inoperability whether distant metastasis or invasive tumours, Patients with synchronous colorectal tumours, synchronous liver metastasis obstructive symptomatic patients and patients with intraoperative tumour rupture or perforation, rectal tumours below peritoneal reflection

Ages: 26 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2016-12-11 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
recovery time-intraoperative bleeding | up to 3 years
Incidence of wound infection | up to 3 years
hospital stay-perioperative length | up to 3 years
oncological outcome | 3 years
  total mesorectal excision, margin included or not

SECONDARY OUTCOMES:
early locoregional recurrence | 6 months
  early locoregional recurrence within 6 months

IPD SHARING:
Plan to Share IPD: Yes
through international publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year
Access Criteria: laparoscopic anterior resection for upper rectal cancer in obese patients

REFERENCES:
- [Result] Kinlen D, Cody D, O'Shea D. Complications of obesity. QJM. 2018 Jul 1;111(7):437-443. doi: 10.1093/qjmed/hcx152. PMID 29025162
- [Result] Allaix ME, Furnee E, Esposito L, Mistrangelo M, Rebecchi F, Arezzo A, Morino M. Analysis of Early and Long-Term Oncologic Outcomes After Converted Laparoscopic Resection Compared to Primary Open Surgery for Rectal Cancer. World J Surg. 2018 Oct;42(10):3405-3414. doi: 10.1007/s00268-018-4614-x. PMID 29610930
- See also: Total Laparoscopic Approach for Rectal Cancer Resection-a Novel Technique and Review of the Literature — https://link.springer.com/article/10.1007/s12262-020-02299-4